CLINICAL TRIAL: NCT02841358
Title: Study Qbout the Screening of Niemann-Pick Disease, Type C in a Psychiatric Population
Brief Title: Screening of Niemann-Pick Disease, Type C in a Psychiatric Population
Acronym: NPCPsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 38RC13.200
Record Dates: First submitted 2016-07-11; First posted 2016-07-22 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Psychiatric Adults Patients
Keywords: Niemann-Pick Disease, Type C; Psychiatric; Psychotic disorders
MeSH Terms: conditions — Niemann-Pick Disease, Type C; Psychotic Disorders | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychiatric adults patients presenting psychologic disorders (Other)
  Interventions: Biological: Blood sampling; Biological: Biopsy

INTERVENTIONS:
Biological: Blood sampling
Biological: Biopsy

SUMMARY:
Niemann-Pick disease, Type C is a rare genetic disorder characterized by a failing in intracellular cholesterol transport, inducing an accumulation of sphingolipids in the brain.

Neurological signs are at the forefront of the disease. There are also psychiatric signs of psychotic kind among 28 to 45 % of patients according to studies, and a thirty cases were published. These signs can be concomitant with neurological signs or precede them.

Is is likely that psychotic disorders are the first signs of a Niemann-Pick disease not yet non encore diagnosed for some patients. Yet, no prevalence study for this disease in a psychiatric population of patients currently exists. In response to this problem this study proposes to search patients whose disease could be of organic origin or patients whose disease is suspected, based on clinical data. The diagnosis will be confirmed certified with a genetic and/or biochemical test.

DETAILED DESCRIPTION:
The aim of this study is to search among a population psychotic adult patients, the ones that present a Type C Niemann-Pick disease in order to to estimate the prevalence.

ELIGIBILITY:
Inclusion Criteria:

* Hallucinations visual
* Confusion
* Catatonia
* Significant fluctuation of symptoms
* Unusual or paradoxical reaction to the treatment
* Progressive cognitive deterioration

Exclusion Criteria:

* Patients under 18 years
* Patients unable to give their free consent and without a legal representative
* Breastfeeding or pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-12; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Blood sampling | 3 minutes
  For patients with suspicion of Type C Niemann-Pick Disease, to determine blood/plasma oxysterols level.
Blood sampling | 2 to 4 half days
  For patients with no longer suspicion of Type C Niemann-Pick Disease, according to blood/plasma oxysterols level, for genotyping with the search of NPC 1 or NPC 2 mutation.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Buis, Doctor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Vanier MT. Niemann-Pick disease type C. Orphanet J Rare Dis. 2010 Jun 3;5:16. doi: 10.1186/1750-1172-5-16. PMID 20525256
- [Background] NP-C Guidelines Working Group; Wraith JE, Baumgartner MR, Bembi B, Covanis A, Levade T, Mengel E, Pineda M, Sedel F, Topcu M, Vanier MT, Widner H, Wijburg FA, Patterson MC. Recommendations on the diagnosis and management of Niemann-Pick disease type C. Mol Genet Metab. 2009 Sep-Oct;98(1-2):152-65. doi: 10.1016/j.ymgme.2009.06.008. Epub 2009 Jun 14. PMID 19647672
- [Background] Garver WS, Francis GA, Jelinek D, Shepherd G, Flynn J, Castro G, Walsh Vockley C, Coppock DL, Pettit KM, Heidenreich RA, Meaney FJ. The National Niemann-Pick C1 disease database: report of clinical features and health problems. Am J Med Genet A. 2007 Jun 1;143A(11):1204-11. doi: 10.1002/ajmg.a.31735. PMID 17497724
- [Background] Sevin M, Lesca G, Baumann N, Millat G, Lyon-Caen O, Vanier MT, Sedel F. The adult form of Niemann-Pick disease type C. Brain. 2007 Jan;130(Pt 1):120-33. doi: 10.1093/brain/awl260. Epub 2006 Sep 26. PMID 17003072
- [Background] Webber D, Klünemann H Psychiatric manifestations of Niemann-Pick Disease European Psychiatric Review, 2011;4(1):25-31
- [Background] Walterfang M, Fietz M, Abel L, Bowman E, Mocellin R, Velakoulis D. Gender dimorphism in siblings with schizophrenia-like psychosis due to Niemann-Pick disease type C. J Inherit Metab Dis. 2009 Dec;32 Suppl 1:S221-6. doi: 10.1007/s10545-009-1173-1. Epub 2009 Jul 17. PMID 19609713
- [Background] Sandu S, Jackowski-Dohrmann S, Ladner A, Haberhausen M, Bachmann C. Niemann-Pick disease type C1 presenting with psychosis in an adolescent male. Eur Child Adolesc Psychiatry. 2009 Sep;18(9):583-5. doi: 10.1007/s00787-009-0010-2. Epub 2009 Mar 7. PMID 19267177
- [Background] Trendelenburg G, Vanier MT, Maza S, Millat G, Bohner G, Munz DL, Zschenderlein R. Niemann-Pick type C disease in a 68-year-old patient. J Neurol Neurosurg Psychiatry. 2006 Aug;77(8):997-8. doi: 10.1136/jnnp.2005.086785. No abstract available. PMID 16844962
- [Background] Walterfang M, Fietz M, Fahey M, Sullivan D, Leane P, Lubman DI, Velakoulis D. The neuropsychiatry of Niemann-Pick type C disease in adulthood. J Neuropsychiatry Clin Neurosci. 2006 Spring;18(2):158-70. doi: 10.1176/jnp.2006.18.2.158. PMID 16720792
- [Background] Tyvaert L, Stojkovic T, Cuisset JM, Vanier MT, Turpin JC, De Seze J, Vermersch P. [Presentation of Niemann-Pick type C disease with psychiatric disturbance in an adult]. Rev Neurol (Paris). 2005 Mar;161(3):318-22. doi: 10.1016/s0035-3787(05)85038-6. French. PMID 15800453
- [Background] Battisti C, Tarugi P, Dotti MT, De Stefano N, Vattimo A, Chierichetti F, Calandra S, Federico A. Adult onset Niemann-Pick type C disease: A clinical, neuroimaging and molecular genetic study. Mov Disord. 2003 Nov;18(11):1405-9. doi: 10.1002/mds.10541. PMID 14639697
- [Background] Turpin JC, Baumann N. [Presenting psychiatric and cognitive disorders in adult neurolipidoses]. Rev Neurol (Paris). 2003 Jul;159(6-7 Pt 1):637-47. French. PMID 12910071
- [Background] Josephs KA, Van Gerpen MW, Van Gerpen JA. Adult onset Niemann-Pick disease type C presenting with psychosis. J Neurol Neurosurg Psychiatry. 2003 Apr;74(4):528-9. doi: 10.1136/jnnp.74.4.528. PMID 12640083
- [Background] Imrie J, Vijayaraghaven S, Whitehouse C, Harris S, Heptinstall L, Church H, Cooper A, Besley GT, Wraith JE. Niemann-Pick disease type C in adults. J Inherit Metab Dis. 2002 Oct;25(6):491-500. doi: 10.1023/a:1021259403196. PMID 12555942
- [Background] Campo JV, Stowe R, Slomka G, Byler D, Gracious B. Psychosis as a presentation of physical disease in adolescence: a case of Niemann-Pick disease, type C. Dev Med Child Neurol. 1998 Feb;40(2):126-9. doi: 10.1111/j.1469-8749.1998.tb15374.x. PMID 9489503
- [Background] Shulman LM, David NJ, Weiner WJ. Psychosis as the initial manifestation of adult-onset Niemann-Pick disease type C. Neurology. 1995 Sep;45(9):1739-43. doi: 10.1212/wnl.45.9.1739. PMID 7675237
- [Background] Shulman LM, Lang AE, Jankovic J, David NJ, Weiner WJ. Case 1, 1995: psychosis, dementia, chorea, ataxia, and supranuclear gaze dysfunction. Mov Disord. 1995 May;10(3):257-62. doi: 10.1002/mds.870100304. No abstract available. PMID 7651440
- [Background] Hulette CM, Earl NL, Anthony DC, Crain BJ. Adult onset Niemann-Pick disease type C presenting with dementia and absent organomegaly. Clin Neuropathol. 1992 Nov-Dec;11(6):293-7. PMID 1473312
- [Background] Bonnot O, Leroy A, Lucanto R, Cohen D Pourquoi s'intéresser à la maladie de Niemann-Pick de type C quand on est psychiatre d'enfant et d'adolescent Neuropsychiatrie de l'enfance et de l'adolescence 2011
- [Background] Bonnot O, Cohen D. [Psychiatric and cognitive signs associated with inborn errors of metabolism]. Rev Neurol (Paris). 2011 Dec;167(12):881-5. doi: 10.1016/j.neurol.2011.03.014. Epub 2011 Oct 29. French. PMID 22041824
- [Background] Muller A, Balding DJ, Kluenemann HH, Linden D, Ory DS, Patterson MC, Pineda M, Priller J, Sedel F, Chadha-Boreham H, Wraith JE, Bauer P. Challenges in screening rare diseases: the ZOOM experience. Abstract accepté pour un poster au 28ème congrès de l'" International Society for Pharmacoepidemiology " Barcelone - août 2012" + données internes
- [Background] American Psychiatric Association - DSM IV TR, Manuel diagnostique et statistique des troubles mentaux, 4° édition, Texte révisé (Washington DC, 2000), Traduction française par J-D Guelfi et al., Masson, Paris, 2003, 1120 p.